CLINICAL TRIAL: NCT04074811
Title: Exploring the Feasibility and Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) in a Healthy Population
Brief Title: Feasibility and Efficacy of rTMS in Healthy Persons
Acronym: TPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor and Associate Department Chair, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TPD-1
Record Dates: First submitted 2019-08-20; First posted 2019-08-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Executive Dysfunction; Pain; Mood
MeSH Terms: conditions — Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This pilot study will use a single-blind, left dorsolateral prefrontal cortex (10-Hz) vs. sham, 2-session, within-subjects randomized crossover design.
Who Masked: Participant
Masking Description: Participants will be blinded to the use of active vs. sham rTMS. For the sham condition, the investigators will use a placebo figure-of-8 coil, which looks identical to the active coil, allows the same scalp placement, and produces the same auditory and tactile sensations as active stimulation without affecting cortical excitability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham rTMS (Sham Comparator): Sham rTMS will be applied over the left dorsolateral prefrontal cortex using a sham figure of 8 coil (within-subject crossover). Sham rTMS will consist of the same auditory and tactile stimuli as the active condition, but does not induce an electromagnetic field and does not affect cortical excitability.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Active rTMS (Active Comparator): Active rTMS will be applied over the left dorsolateral prefrontal cortex using an active figure of 8 coil (within-subject crossover). In the active rTMS condition, the investigators will use high-frequency (10Hz) dorsolateral prefrontal cortex (dlPFC) stimulation with intensity of 110% of resting motor threshold. rTMS will consist of 120 trains with 50 stimuli per train (i.e. 5-sec long at 10 Hz) and 10-sec intertrain interval for a total of 6000 pulses. The entire protocol will last 30 min (120 trains with 5-sec on/10-sec off).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — The investigators will use the Figure of 8 coil, which affects ~10cm2 of cortical surface. The active condition will deliver stimulation at 110% of resting motor threshold (RMT). To determine RMT, the protocol will be: 10 trials of single-pulse TMS on the scalp position of the abductor pollicis brevis muscle (which controls thumb flexion); RMT is the lowest TMS power setting yielding visible motor contraction on >50% of trials.

SUMMARY:
Transcranial magnetic stimulation (TMS) is a neuromodulation device that is FDA-approved for use in treating depression and obsessive compulsive disorder. TMS works by applying a safe, electromagnetic field on the scalp, which can either increase or decrease neuronal communication and activity (depending on the mode of stimulation). Although it is only approved for two disorders, there has been substantial research into the potential of TMS to treat a wide range of neuropsychiatric disorders, including substance use disorders (SUDs). This project aims to develop an initial TMS protocol in a sample of healthy controls and to establish the feasibility and efficacy of using repetitive TMS (rTMS) to impact several carefully-selected cognitive, behavioral, and physiologic measures. This pilot project will enable the research team to gather baseline data using this new method and to plan longer-term programmatic studies focusing on populations with SUDs. The overarching aim of this project is to develop an rTMS protocol for use in the human laboratory setting with both healthy controls and individuals with SUDs. The investigators also hope to learn about the impact of high frequency rTMS over the DLPFC on multiple aspects of functioning including: cognitive control, impulsivity, thermal pain sensitivity, motivation, and mood.

DETAILED DESCRIPTION:
The short-term goal of this pilot project is to establish the feasibility and efficacy of repetitive transcranial magnetic stimulation (rTMS) on cognitive, behavioral, and physiological measures in a healthy community-recruited sample to plan longer-term programmatic studies focusing on substance use disorder (SUD) populations. Primary Aims are to examine the effect of one session of left dorsolateral prefrontal cortex (DLPFC) rTMS high-frequency (10 Hz) stimulation vs. placebo stimulation (no electromagnetic field but similar auditory and tactile sensations) on: (1) cognitive control, (2), impulsivity, and (3) thermal pain sensitivity. Secondary Aims are to test effects of rTMS on behavioral motivation (monetary incentive delay task, effort choice task), mood (PANAS), peripheral biomarkers (prolactin, BDNF) and collect biosamples for future genotyping.

The investigators recognize the proposed sample size is relatively small to adequately power a full analysis across all outcomes, so will use this study to determine effect sizes for any differences to plan future studies with adequate power. Generally speaking, data will be analyzed using repeated measures ANCOVAs; covariates will include TMS resting motor threshold, sex, and age. Based on sample size calculations, the investigators intend to complete up to 30 subjects. For some outcomes, the results of previous studies indicate that a lower sample size may be appropriate, therefore the investigators will conduct interim analyses at n=18 to calculate effect sizes to determine how many more participants are needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Right handed
* 21-60 years of age
* IQ score greater than 80
* Eligible if using tobacco, alcohol, or marijuana fewer than 3 times per week; each "time" must be less than 3 cigarettes or drinks, or less than 1 marijuana "joint"

Exclusion Criteria:

* Under influence of any substances during any session
* Use of illicit substances in the past 30 days
* Pregnant
* Medical conditions that prohibit the use of rTMS (e.g. history of seizures or medications that lower seizure threshold)
* Current DSM-5 Axis I psychiatric disorders, or any history of substance use disorders.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Stroop Task (cognitive control) | Change from pre- to 25-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on cognitive control as measured by the Stroop Color-Word task.
Stop Signal Task (impulsivity) | Change from pre- to 15-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on impulsivity as measured by the Stop Signal Task.
Pain Sensitivity | Change from pre- to 50-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on pain sensitivity as measured by thermal quantitative sensory threshold (QST) testing.
Delay Discounting Task (cognitive control) | Change from pre- to 10-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on cognitive control as measured by the brief (2-min) monetary delay discounting task

SECONDARY OUTCOMES:
Effort Choice Task (motivation) | Change from pre- to 30-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on behavioral responding as measured by the Effort Choice Task (number of responses on progressive ratio vs. fixed ratio schedules of reinforcement).
Mood | Change from pre- to 5-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on mood state as measured by the Positive and Negative Affect Schedule.
Peripheral Biomarkers | Change from pre- to 0-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on peripheral biomarkers as measured by the plasma concentrations (ng/ml) of brain derived neurotrophic factor (BDNF) and prolactin.
Monetary Incentive Delay Task (motivation) | Change from pre- to 40-minutes post-rTMS stimulation in each session
  Examine the effect of rTMS stimulation on behavioral responding as measured by the Monetary Incentive Delay Task

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team is committed to disclosing and sharing scientific findings as outlined by NIH policy guidance on Sharing Research Data and on Sharing Model Organisms (see: http://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm#time). We note that, "NIH recognizes that the investigators who collected the data have a legitimate interest in benefiting from their investment of time and effort. NIH continues to expect that the initial investigators may benefit from first and continuing use but not from prolonged exclusive use." The research team (PI, with advice from co-investigators) plans to share data from this project as follows. We will disseminate data using conventional means including published abstracts, conference presentations (posters and talks), news releases, and peer reviewed journal articles.
Supporting Information: CSR
Time Frame: Findings from the proposed investigation will be provided to the scientific community as rapidly as possible, given the usual constraints of careful data checking, analysis, and peer review.
Access Criteria: Qualified researchers may request in writing additional protocol materials from the PI.